CLINICAL TRIAL: NCT05750199
Title: The Effectiveness of "Multi-Immunotherapy Special Training Courses Through Digital Media and Workshop" Intervention for Oncology Nurses: Exploration of Educational Needs, Curriculum Planning, Implementation and Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201912255RINC
Record Dates: First submitted 2022-01-06; First posted 2023-03-01 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Education; Oncology; Immune
Keywords: cancer; immunotherapy; oncology nurse; education need; training course
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immunotherapy Special Training Course (ISTC) (Experimental): 16 weeks and includes 8 hours of digital media training and 2 days of workshop training.
  Interventions: Other: Immunotherapy Special Training Course (ISTC)
- Advanced Oncology Nurse Training Course (AONTC) (Experimental): 4 weeks and includes 8 days of Advanced Oncology Nurse Training Course.
  Interventions: Other: Advanced Oncology Nurse Training Course (AONTC)

INTERVENTIONS:
Other: Immunotherapy Special Training Course (ISTC) — 16 weeks and includes 8 hours of digital media training and 2 days of workshop training.
  Arms: Immunotherapy Special Training Course (ISTC)
Other: Advanced Oncology Nurse Training Course (AONTC) — 4 weeks and includes 8 days of Advanced Oncology Nurse Training Course
  Arms: Advanced Oncology Nurse Training Course (AONTC)

SUMMARY:
This study is a 2-year qualitative and quantitative mixed method research project and consists of two phases.The study will provide useful clinical data to help us better understand educational needs of immunotherapy for oncology nurses. This ISTC model will lead to further validation of an oncology care training course model designed to better prepare and support cancer patients and their families to existing and new anti-cancer therapies.

DETAILED DESCRIPTION:
Background: More and more cancer patients are receiving immunotherapy. However, patients and their families are overwhelmingly not fully aware of the side effects of immunotherapy or the related management involved while simultaneously experiencing both financial and spiritual burden. Thus, educating the needs of immunotherapy and the development and planning of immunotherapy-related training courses for oncology nurses are necessary.

Purpose: (1) To explore the educational needs for immunotherapy in oncology nurses. (2) To develop and evaluate the effectiveness of "Multi-Immunotherapy Special Training Courses through Digital Media and Workshop" intervention" (short for Immunotherapy Special Training Course (ISTC)" on immunotherapy related care indicators and the feasibility of the ISTC.

Method: This study is a 2-year qualitative and quantitative mixed method research project and consists of two phases: (1) The qualitative method will be conducted using phenomenological methods and snowball sampling. In-depth interviews and observations by one researcher will be adopted in this study. The sample size is determined as the number of samples collected until saturated data analysis is achieved. (2) The quantitative method will be conducted as a quasi-experimental research with a two group pretest-posttest. For the experimental group, snowball sampling will be used to recruit participants who are recommended by a cooperative teaching hospital in the North, Central, South and East Districts of Taiwan to participate in the ISTC training. The duration is to last 16 weeks and includes 8 hours of digital media training and 2 days of workshop training. For the control group, convenient sampling will be used to recruit participants attending the "Advanced Oncology Nurse Training Course (AONTC) (during 4 weeks, 8 days)." which will be held by the Taiwan Oncology Nursing Society. Each group will be followed for 3 to 4 months and their outcomes will be assessed at 3 time points: baseline (pre-training course), and 8, 12 weeks after the training course, T0-T2, respectively. Outcomes will be evaluated based on immunotherapy knowledge, self-efficacy of caring responsible for patients undergoing immunotherapy, critical thinking ability, and ability of communication. Additionally, in the experimental group, outcomes will also be evaluated by mini-clinical evaluation exercise, mini-CEX at T2 and learning passport at 16 weeks after training course (T3). Estimated subject number would be 60 for each group. Results would be analyzed mainly by GEE. After obtaining approval from the institutional review board of a medical center in northern Taiwan and getting the required consent, this study will commence.

Predicted results: The study will provide useful clinical data to help us better understand educational needs of immunotherapy for oncology nurses. This ISTC model will lead to further validation of an oncology care training course model designed to better prepare and support cancer patients and their families to existing and new anti-cancer therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Over 20 years old (inclusive).
2. Nurses or case managers who have completed the training of oncology nursing courses in their hospitals.
3. Caring experiences of cancer patients who undergoing immunotherapy.
4. The working experience of the oncology unit is at least 1 years.

Exclusion Criteria:

1. Those who are unwilling or unable to participate in the full four-month course training.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
Educational needs | 1 time points:first time is before the training course
  Oncology nurses' educational needs for immunotherapy will be assesed qualitative method.

SECONDARY OUTCOMES:
Communication ability scale | 2 time points: Time 1 (before the training course) ; Time 2 (16 weeks after the training course)
  Oncology nurses' communication skills were measured by communication ability scale.It is a 5 Liker scale(1-5),higher scores represent better communication skills
Self efficacy scale | 2 time points: Time 1 (before the training course) ; Time 2 (16 weeks after the training course)
  Oncology nurses' self efficacy will measure by Self efficacy scale.It is a 11 point (0-10) scale.The higher the score, the more confident you are in caring for immunotherapy patients or their families.
Critical Thinking test | 2 time points: Time 1 (before the training course) ; Time 2 (16 weeks after the training course)
  Effects of oncology nurses received immunization course will measure by Critical Thinking test .It is a 6 Liker scale (1-6) ,the higher score indicates that the participant the better the ability to think critically.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University, Taipei, Taiwan